CLINICAL TRIAL: NCT00713739
Title: Evaluation of Alfuzosin as Medical Expulsion Therapy for Ureteral Stones
Brief Title: Alfuzosin for Medical Expulsion Therapy of Ureteral Stones
Acronym: MET
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Responsible Party: Principal Investigator, Sean Stroup, Principle Investigator, United States Naval Medical Center, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMCSD CID 06-050; Office of Naval Research FY08
Record Dates: First submitted 2008-07-07; First posted 2008-07-11 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Kidney Stones
Keywords: kidney stones; ureteral stones; medical expulsion therapy
MeSH Terms: conditions — Kidney Calculi | interventions — alfuzosin; Nifedipine; Doxazosin; Prazosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Alfuzosin 10mg daily
  Interventions: Drug: Alfuzosin
- 2 (Active Comparator): Nifedipine XL 30mg daily
  Interventions: Drug: nifedipine
- 3 (Active Comparator): Doxazosin 4 mg daily
  Interventions: Drug: doxazosin
- 4 (Active Comparator): Prazosin 1 mg BID
  Interventions: Drug: prazosin

INTERVENTIONS:
Drug: Alfuzosin — Patients who present to NMCSD with symptomatic ureteral stones visible on CT and KUB, and who are medically stable will be offered enrollment. The patients will be randomly assigned to one of 4 groups. Outpatient treatment groups will be randomized 1:1:1:1 and include; Group 1 - Alfuzosin 10 mg daily, Group 2 - Nifedipine 30 mg daily, Group 3 - Doxazosin 4 mg daily, or Group 4 - Prazosin 1 mg BID. The treatment regimens consist of daily medication until the stone passes or 21 days, whatever is shorter. Patients will also receive oral pain medication as needed.
  Arms: 1
Drug: nifedipine — Patients who present to NMCSD with symptomatic ureteral stones visible on CT and KUB, and who are medically stable will be offered enrollment. The patients will be randomly assigned to one of 4 groups. Outpatient treatment groups will be randomized 1:1:1:1 and include; Group 1 - Alfuzosin 10 mg daily, Group 2 - Nifedipine 30 mg daily, Group 3 - Doxazosin 4 mg daily, or Group 4 - Prazosin 1 mg BID. The treatment regimens consist of daily medication until the stone passes or 21 days, whatever is shorter. Patients will also receive oral pain medication as needed.
  Arms: 2
Drug: doxazosin — Patients who present to NMCSD with symptomatic ureteral stones visible on CT and KUB, and who are medically stable will be offered enrollment. The patients will be randomly assigned to one of 4 groups. Outpatient treatment groups will be randomized 1:1:1:1 and include; Group 1 - Alfuzosin 10 mg daily, Group 2 - Nifedipine 30 mg daily, Group 3 - Doxazosin 4 mg daily, or Group 4 - Prazosin 1 mg BID. The treatment regimens consist of daily medication until the stone passes or 21 days, whatever is shorter. Patients will also receive oral pain medication as needed.
  Arms: 3
Drug: prazosin — Patients who present to NMCSD with symptomatic ureteral stones visible on CT and KUB, and who are medically stable will be offered enrollment. The patients will be randomly assigned to one of 4 groups. Outpatient treatment groups will be randomized 1:1:1:1 and include; Group 1 - Alfuzosin 10 mg daily, Group 2 - Nifedipine 30 mg daily, Group 3 - Doxazosin 4 mg daily, or Group 4 - Prazosin 1 mg BID. The treatment regimens consist of daily medication until the stone passes or 21 days, whatever is shorter. Patients will also receive oral pain medication as needed.
  Arms: 4

SUMMARY:
The goal of this study is to conduct a prospective controlled trail of four currently approved Department of Defense (DOD) - formulary medications for use as medical expulsion therapy (MET) for kidney stones. Between 8% and 15% of Americans will develop symptomatic urolithiasis in there life. Several medications, including steroids, calcium channel blockers, alpha-adrenergic antagonists and non-steroidal anti-inflammatory drugs, have been utilized to aid in the spontaneous passage of distal ureteral calculi. Recently, use of selective alpha-blockers has shown promise for medical expulsion therapy (MET) of distal ureteral calculi. None of these studies have been widely publicized outside the specialty of urology. Recent studies have shown a success rate of nearly 90% when the selective alpha-blocker tamsulosin (Flomax) was used for MET. MET has also been shown to result in a decreased narcotic requirement, shorter time to stone passage, and reduced requirement for further interventions. The investigators will evaluate the effectiveness of MET as initial management for kidney stones using DOD-approved formulary medications.

DETAILED DESCRIPTION:
Patients presenting to Naval Medical Center San Diego with symptomatic ureteral stones visible on CT and KUB, and who are medically stable will be offered enrollment. Upon consent, patients will be randomly assigned to one of four outpatient treatment arms, randomized 1:1:1:1 and include; Group 1 - Alfuzosin 10 mg daily, Group 2 - Nifedipine 30 mg daily, Group 3 - Doxazosin 4 mg daily, or Group 4 - Prazosin 1 mg twice daily. The primary endpoint is stone expulsion rate and secondary endpoints are time to expulsion, need for additional intervention, degree of pain control, amount of narcotic use, and evaluation of study drug side effects. The treatment regimens consist of daily medication until the stone passes or 21 days, whatever is shorter. Patients will also receive oral pain medication as needed.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18 years
* Single ureteral stone < 1 cm in greatest dimension

Exclusion Criteria:

* Age < 18 years
* Active unstable angina
* History of or active postural hypotension (>20 mmHg drop in orthostatic SBP)
* Allergy to alpha-blockers
* Acute or Chronic Renal Failure as demonstrated by a serum creatinine of > 1.4 mg/dl
* Urinary tract infection
* Multiple ureteral stones
* Current uncontrolled diabetes
* Alpha-blocker therapy within 30 days for any reason
* Current pregnancy or lactation
* Patient desire for immediate stone removal

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2008-01; Primary Completion 2010-12 (Actual); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
The primary measures are percent of stones passed and rates of occurrence of various side effects (categorical variables), and time to pass, pain scale, and amount of pain medication taken (continuous variables). | Period of stone passage (30 days)

CONTACTS AND LOCATIONS:
Overall Officials: Brian K. Auge, M.D., Principal Investigator — NMCSD; Sean P. Stroup, M.D., Principal Investigator — NMCSD
Locations (1):
- Naval Medical Center San Diego, San Diego, California, United States